CLINICAL TRIAL: NCT05521542
Title: ADVANCEd NanoTherapies Dual Active Pharmacological Ingredient (Dual-API) Drug-Coated Balloon Catheter to Treat De-Novo Lesions in Patients With Symptomatic Stable Angina, Unstable Angina, and NSTEMI
Brief Title: Advanced NanoTherapies Dual-API DCB to Treat De-Novo Lesions in Patients With Symptomatic Coronary Artery Disease
Acronym: ADVANCE-DCB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced NanoTherapies (Industry)
Collaborators: Monash University (Other); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDNV-001
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: Drug Coated Ballon; DCB; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single-arm, feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SirPlux™ Duo Dual-API Coated PTCA Balloon Catheter (Experimental): Subjects who meet the inclusion criteria and agree to participate in the study will be enrolled and undergo a planned percutaneous coronary intervention with SirPlux™.
  Interventions: Device: SirPlux Duo™ Dual-API Coated PTCA Balloon Catheter

INTERVENTIONS:
Device: SirPlux Duo™ Dual-API Coated PTCA Balloon Catheter — SirPlux Duo™ Dual-API Coated PTCA Balloon Catheter is a Drug-Coated Balloon to treat de novo lesions in patients with symptomatic stable angina, unstable angina, or NSTEMI

SUMMARY:
This prospective, single-arm, multi-center, safety and feasibility first-in-human study will evaluate the safety and feasibility of the SirPlux Duo™ Dual-API Coated PTCA Balloon Catheter to treat de-novo lesions between ≥2.0 and ≤4.0 mm in patients with symptomatic stable angina, unstable angina, and NSTEMI.

DETAILED DESCRIPTION:
The SirPlux Duo™ Dual API-Coated PTCA Balloon Catheter is an investigational medical device to be used to treat de-novo lesions in patients with symptomatic stable angina, unstable angina, and NSTEMI. In this study, SirPlux Duo™ will be used in subjects undergoing a planned percutaneous coronary intervention. The population to treat will include those with de-novo coronary lesions in vessels with a reference vessel diameter (RVD) of ≥2.0 and ≤4.0 mm and a total lesion length of <36mm with documented symptomatic stable angina, unstable angina, or NSTEMI. The study is a prospective, single-arm, multi-center, safety and feasibility first-in-human study designed to generate descriptive data about the use of SirPlux Duo™.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is ≥18 years and <90 years old.
2. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed.
3. Subject has been diagnosed with a symptomatic stable angina, or acute coronary syndrome.
4. Life expectancy > 1 year.
5. The subject is planned to undergo a percutaneous coronary intervention for a known lesion meeting the angiographic criteria set out below.
6. Women of child-bearing potential must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure. Men with a female partner of childbearing potential must agree to use condoms plus an additional reliable contraceptive method within 12 months after the index procedure.
7. The subject is able and willing to comply with all assessments in the study, including dual antiplatelet therapy (DAPT), ASA indefinitely, and P2Y12 inhibitor for a minimum of 6 months for stable angina subjects, and 12 months for unstable angina and NSTEMI subjects.
8. The subject shall be under optimal medical therapy for ASCVD, which includes at a minimum high-intensity statin therapy. If statin intolerant, the subject should be treated with a PCSK9 inhibitor, ezetimibe or bempedoic acid.

   Angiographic Inclusion Criteria:
9. Target lesion is located within a de-novo lesion located in a native coronary artery with a reference vessel diameter between and including 2.0 mm and 4.0mm by visual estimate, with an in-segment length <=36mm. Target lesions must have a visually estimated stenosis of ≥50% and be <100% in symptomatic subjects prior to lesion pre-dilation.
10. Subject has one or two lesions that meet inclusion and exclusion criteria individually that could be treated with a study device.

    If multiple lesions are treated, only two may be treated with the investigational device.

    If two lesions are treated with the investigational device, they must be in different vessels.

    Non-target lesions (lesion to be treated with something other than the investigational device) may be treated at either baseline or staged PCI but never in the same vessel as the target lesion.
11. Successful pre-dilation with semi and/or non-compliant balloon of the target lesion(s) (defined as no major flow-limiting dissections (Grade C or higher) and <30% residual stenosis of the target lesion by a visual estimate on angiography). Adjunctive pre-dilation therapies such as scoring balloon, cutting balloon, and IVL are allowed. Rotablator or similar rotational atherectomy devices are restricted per protocol.

Exclusion Criteria:

General Exclusion Criteria:

1. Subject has current problems with substance abuse.
2. Subject has a planned procedure that may cause non-compliance with the protocol.
3. Subject participates in another investigational drug or device clinical study that has not reached its primary endpoint.
4. Subject intends to participate in another investigational drug or device clinical study within 12 months after the index procedure.
5. Chronic total occlusion (CTO) of the target lesion(s) or Thrombolysis In Myocardial Infarction (TIMI) flow < 2.
6. Subject requires treatment of a coronary lesion(s) involving a bifurcation with significant ostial / proximal disease within 5mm of a side-branch greater than 2.0mm.
7. Target lesion(s) within native or synthetic vessel grafts.
8. Subject has had any major (e.g., cardiac, and non-cardiac) surgical procedure or intervention unrelated to this study within 30 days before the index procedure or has a planned major surgical procedure or intervention within 30 days of the index procedure. The exception will be made in case of planned staged PCI procedures for other coronary lesions (study or non-study lesion) lesions, whereby the timeframe between procedures shall be determined by the clinical stability of the subject as assessed by the treating investigator. The subject must re-meet the inclusion criteria and be free from any exclusion criteria before enrolment.
9. The subject has a known coagulopathy or has a bleeding diathesis, thrombocytopenia (with platelet counts less than 100,000/microliter) or platelets > 450,000/microliter, or international normalized ratio >1.5. Subjects on chronic oral anticoagulation medications will be excluded of the study.
10. Known renal insufficiency, estimated glomerular filtration rate (eGFR) ≤30 mL/min, by institutional calculation.
11. Subject on dialysis, or acute kidney failure (as per physician judgment).
12. Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated or hypersensitive.
13. Subject has a known allergy to contrast agents or medications used to perform a coronary intervention that cannot be adequately pre-treated, including, but not limited to, sirolimus, paclitaxel, aspirin, heparin, clopidogrel bisulfate, ticlopidine, prasugrel, ticagrelor.
14. Subject has a known allergy to urethane, nylon, or silicone.
15. Presentation and index admission with STEMI. An exception to this exclusion is the treatment of the non-culprit target lesion with study device during a staged PCI procedure which can be either during the index STEMI admission (but not at the time of primary PCI) or electively at another date.
16. Type 2 NSTEMI
17. Presentation with ACS and ongoing chest pain and/or hemodynamic instability despite treatment of the culprit lesion
18. History of stroke/TIA within 60 days before enrollment.
19. LVEF less than or equal to 35%.
20. Subject is confined to bed.
21. History of thrombolytic therapy within two weeks of enrollment.
22. Subject is a recipient of a heart transplant.
23. Subject is unwilling/not able to return for angiographic catheterization at 6-month follow-up.
24. Women who are pregnant, breast-feeding or intend to become pregnant.
25. Subject has other medical, social, or psychological problems and is unwilling or unable to comply with procedures specified in the protocol or may have difficulty returning for follow-up visits as specified by the protocol.
26. Cardiogenic shock (SBP <80mmHg requiring inotropes, IABP, or fluid support).
27. Subject has symptomatic active COVID-19 or is asymptomatic within the past 2 weeks of a positive COVID test.

    Angiographic Exclusion Criteria:
28. Subject has a planned intervention in the left-main plus two separate major epicardial territories (left-main plus 2 vessel diseases).
29. Target vessel size <2.00 mm or >4.0 mm
30. Target lesion in the left main stem.
31. Target vessel with high thrombus burden.
32. Aorto-ostial target RCA lesion (within < 10 mm of the aorta junction)
33. Moderate-severe tortuous, calcified, or angulated coronary anatomy of the target vessel that, in the opinion of the Investigator, would result in suboptimal imaging or excessive risk of complication from placement of an IVUS catheter following Clinical Decision.
34. The lesion is located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft.
35. Target lesion is located within a previous implanted stent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Device Success | (Peri-procedural)
  Defined as successful delivery, balloon inflation, deflation, and retrieval of the intact study device without burst below rated burst pressure
Technical Success | (Peri-procedural)
  Defined as successful lesion crossing, completion of POBA and immediate achievement of <=30% residual stenosis (by QCA) of the target lesion upon completion of angiography post investigational device inflation
Procedural Success | (Peri-procedural)
  Defined as device success and technical success and absence of procedural complications following SirPlux Duo™ Dual-API Coated PTCA Balloon Catheter inflation (ie absence of vessel dissection or loss of TIMI 3 flow)
In-segment Late Lumen Loss (LLL) by QCA | 6 months post-procedure
  difference in minimum lumen diameter, as determined by QCA, from baseline (immediately post-DCB) to 6 months post-procedure

SECONDARY OUTCOMES:
All-cause death | 24 hours post-discharge
  All-cause death, including death during procedure and up to 24 hours after discharge
  * Target Vessel Myocardial Infarction (TVMI).
  * Cardiac death
  * Myocardial Infarction (MI)
  * Emergent Coronary Artery Bypass Graft (CABG)
  * Repeat Target Lesion Revascularization (TLR) (clinically driven) by percutaneous or surgical methods
  * Major Adverse Cardiac Event (MACE)
  * Target Vessel Failure (TVF)
  * Target Lesion Failure (TLF)
  * All revascularizations (TLR, TVR and non-TVR)
Target Vessel Myocardial Infarction (TVMI) | 30 days, 6 months, 12 months and 24 months post-procedure
  • Target Vessel Myocardial Infarction (TVMI)
Major Adverse Cardiac Event (MACE) | 30 days, 6 months, 12 months and 24 months post-procedure
  • Major Adverse Cardiac Event (MACE) is defined as the composite of cardiac death, Myocardial Infarction (MI), emergent Coronary Artery Bypass Graft (CABG), or repeat Target Lesion Revascularization (TLR) (clinically driven) by percutaneous or surgical methods
Target Vessel Failure (TVF) | 30 days, 6 months, 12 months and 24 months post-procedure
  • Target Vessel Failure (TVF) is defined as cardiac death, TVMI, or clinically-driven Target Vessel Revascularization (TVR) by percutaneous or surgical methods of the target vessel
Target Lesion Failure (TLF) | 30 days, 6 months, 12 months and 24 months post-procedure
  • Target Lesion Failure (TLF) is defined by a composite of cardiac death, TVMI, or clinically driven TLR by percutaneous or surgical methods of the index lesion
All revascularizations (TLR, TVR and non-TVR) | 30 days, 6 months, 12 months and 24 months post-procedure
  • All revascularizations (TLR, TVR and non-TVR) as a composite of TLR, TVR, and non-TVR
In-segment (in balloon) percent diameter stenosis (%DS) by QCA | 6 months post-procedure
  In-segment (in balloon) percent diameter stenosis (% diameter stenosis; %DS).
In-segment binary angiographic restenosis (BAR) rate by QCA | 6 months post-procedure
  In-segment binary angiographic restenosis (BAR) is defined as ≥50% diameter stenosis.
In-segment Minimum Luminal/Lumen Diameter (MLD) by QCA | 6 months post-procedure
  In-segment Minimum Luminal/Lumen Diameter (MLD) change from baseline to 6 months post-procedure
In-segment Change in IVUS minimum lumen area (MLA, mm2) by IVUS | at 6 months post-procedure
  In-segment Change in IVUS MLA (mm2) from baseline to 6 months post-procedure
In-segment change in mean lumen area (mm2) by IVUS | 6 months post-procedure
  In-segment change in mean lumen area (mm2) from baseline to 6 months post-procedure
In-segment change in percentage atheroma volume by IVUS | 6 months post-procedure
  In-segment change in percentage atheroma volume from baseline to 6 months post-procedure
In-segment serial IVUS remodeling | 6 months post-procedure
  In-segment Serial IVUS remodeling (change in vessel area or volume) from baseline to 6 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholls, Study Director — Monash Heart
Locations (5):
- Australia (3):
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Victorian Heart Institute - Monash University, Clayton, Victoria
- Cecanot Hospital, Santo Domingo, Dominican Republic
- Te Toka Tumai Auckland, Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No